CLINICAL TRIAL: NCT06032013
Title: Patient-Reported Outcome Measures and Quality of Life in Cardiac Rehabilitation: Impact on Health Care
Brief Title: Patient-Reported Outcome Measures in Cardiac Rehabilitation: Impact on Health Care
Acronym: PROM_R
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed with fewer participants than expected
Sponsor: José Manuel Afonso Moreira (Other)
Responsible Party: Sponsor-Investigator, José Manuel Afonso Moreira, Principal Investigator, University of Évora
Organization: University of Évora (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: National School Public Health
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life; Cardiac Rehabilitation; Patient-Reported Outcome Measures; Rehabilitation Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Rehabilitation intervention (Experimental): Outpatient intervention with participants after a cardiac event who fulfil the inclusion criteria.
  Interventions: Other: Cardiac rehabilitation program (PROMs)

INTERVENTIONS:
Other: Cardiac rehabilitation program (PROMs) — The program is multidisciplinary with the following components:
  * Medical assessment
  * Physical training and counselling on physical activity
  * Identification and control of risk factors
  * Nutritional assessment and counselling
  * Psychological assessment and intervention
  * Education and information

SUMMARY:
Cardiac Rehabilitation (CR) programs are a multidisciplinary process aimed at patient recovery after an acute cardiovascular event or with chronic heart disease, reducing mortality and morbidity, optimising functional capacity and improving quality of life. The aim is to maintain or recover the patient's clinical, physical and psychosocial condition, slowing down or halting the progression of the underlying disease process. It is based on the practice of personalized physical exercise and the adaptation of behaviours towards a healthier lifestyle, ensuring the reduction and control of risk factors. It is considered a cost-effective intervention that is explicitly and formally recommended by the most diverse and important scientific societies. Through the partnership and collaboration between the various health institutions and the academy, the CR program will take place on an outpatient basis, in a supervised manner, starting after risk stratification with a stress test and respective clinical assessment by a cardiologist. The coordinator of the CR program will be a cardiologist, and the entire multidisciplinary team will be responsible for effectiveness and safety, as well as patient assessment and progress.

DETAILED DESCRIPTION:
The outpatient CR program is designed for a group of participants who have had a cardiac event, based on the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription, consisting of two exercise sessions/week. The sessions are supervised by a healthcare professional specialising in cardiac rehabilitation, and the participant's haemodynamic status is monitored continuously using scales and electronic equipment. PROMs will be applied before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years);
* Low-moderate risk for physical exercise;
* After a cardiac event;
* Have signed an informed consent form.

Exclusion Criteria:

* Physical or mental limitation to carry out an exercise programme;
* Uncontrolled arrhythmia;
* Severe chronic obstructive pulmonary disease;
* Uncontrolled hypertension;
* Symptomatic peripheral arterial disease;
* Unstable angina;
* Uncontrolled diabetes;
* Acute pulmonary oedema in the last 12 hours;
* Those who refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L: Health-related quality of life | Before the intervention and up to 8 weeks.
  The EQ5D makes it possible to assess quality of life in a given pathology in the general population, presented in different domains. The visual analogue scale of this questionnaire has a score of 0-100. Higher scores mean a better result.
HADS: Anxiety and depression | Before the intervention and up to 8 weeks.
  Participants' anxiety and worries are also assessed. Mood disorders, weakness, worry, stress, and depression are common psychological repercussions for patients after a cardiac event, which can trigger hyperventilation reactions. This type of common reaction to emotional extremes such as fear, anxiety, or stress in participants can have a direct impact on involvement in CR programs. This questionnaire is made up of 14 questions. Lower scores mean a better result.
BREQ-2: Behavioural Regulations in Exercise Questionnaire | Before the intervention and up to 8 weeks.
  Assessment of the different aspects of motivational regulation for exercise. It is a questionnaire that evaluates and represents the differences in the ways in which people's behaviour can be regulated and how these differences are experienced.

SECONDARY OUTCOMES:
Heart rate | Before, during and up to 8 weeks of the program.
  Heart rate (bpm)
Blood pressure | Before, during and up to 8 weeks of the program.
  Blood pressure (mmHg)
Peripheral oxygen saturation | Before, during and up to 8 weeks of the program.
  Peripheral oxygen saturation (%)
Exercise Capacity | During and up to 8 weeks of the program.
  Borg scale- score 0-10. Higher values mean greater respiratory effort.
Weight | Before the intervention and up to 8 weeks.
  Weight (Kg)
Abdominal perimeter | Before the intervention and up to 8 weeks.
  Abdominal perimeter (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- National School of Public Health, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No